CLINICAL TRIAL: NCT01479231
Title: Predictors of PPI Response in Eosinophilic Esophagitis
Brief Title: Predictors of Proton Pump Inhibitor (PPI) Response in Eosinophilic Esophagitis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Souces of funding have been terminated
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey A Alexander, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-003759
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Gastroesophageal Reflux Disease; Eosinophilic Esophagitis; Dysphagia
Keywords: GERD; Eosinophilic esophagitis; Proton pump inhibitor; dysphagia
MeSH Terms: conditions — Gastroesophageal Reflux; Eosinophilic Esophagitis; Deglutition Disorders | interventions — Dexlansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dexlansoprazole (Experimental)
  Interventions: Drug: dexlansoprazole

INTERVENTIONS:
Drug: dexlansoprazole — Dexlansoprazole 60 mg daily for 6 weeks
  Other Names: Dexilant

SUMMARY:
The investigators will determine the prevalence of gastroesophageal reflux disease (GERD) in Eosinophilic Esophagitis (EoE) and importantly determine the predictors of response to Proton Pump Inhibitor (PPI) therapy in EoE. Moreover, the investigators will determine the effect of GERD on the location of esophageal eosinophilia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age < 80 years of age
* 14 eosinophils / hpf on biopsies from esophagus

  * Abnormal validated Mayo dysphagia questionnaire (MDQ-30) (question 2"yes", question 4 > "moderate" and question 7 > "once a week")
  * Clinically performed EGD with > 14 eosinophils/hpf completed within last 3 months

Exclusion Criteria:

* Other cause of dysphagia identified at endoscopy (e.g. stricture, web, infection, ring, achalasia, esophageal neoplasm)
* Dilatation of esophagus at time of index endoscopy
* Treatment with topical steroid within 3 months of index endoscopy
* Treatment with PPI in last 30 days prior to index EGD

Patient population - adults with EoE recruited from Mayo Clinic Rochester, MN patient population

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of Gastroesophageal Reflux Disease | 24 hour
  Prevalence of Gastroesophageal Reflux Disease (GERD) in Eosinophilic Esophagitis (EoE) Description: The definition of GERD is acid exposure time of >4.2% over 24 hour period, as measured by pH monitoring.

SECONDARY OUTCOMES:
Heartburn/regurgitation | 30 day
  Heartburn/regurgitation (as measured by:) Mayo Dysphagia Questionnaire - 30 Day Validated 28 item instrument; 0 = no dysphagia, higher levels indicate greater dysphagia severity. Dysphagia. 2010 Sep;25(3):221-30 Measured by "units on a scale"
Abnormal 24 hour acid exposure | 24 hour
  Abnormal 24 hour acid exposure (as measured by pH monitoring) Description: A thin plastic catheter is passed through one nostril, down the back of the throat, and into the esophagus as the patient swallows. The tip of the catheter contains a sensor that senses acid. The catheter protruding from the nose is connected to a recorder that registers each reflux of acid. The catheter is in place for 24 hours, when is removed and the recorder is attached to a computer so that the data can be downloaded.
Ratio of distal/proximal mean esophageal eosinophil number | 6 weeks
  Ratio of distal/proximal mean esophageal eosinophil number (as measured by biopsies taken during esophagogastroduodenoscopy (EGD))
Mean distal eosinophil number | 6 weeks
  Mean distal eosinophil number (as measured by biopsies taken during esophagogastroduodenoscopy (EGD) )

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Alexander, MD, Principal Investigator — Mayo Clinic